CLINICAL TRIAL: NCT02733913
Title: Clinical Impact of Autonomic Modulation After Pulmonary Vein Isolation in Patients With Paroxysmal Atrial Fibrillation
Brief Title: Clinical Impact of Autonomic Modulation After Pulmonary Vein Isolation
Status: Completed | Type: Observational
Sponsor: Klinik für Kardiologie, Pneumologie und Angiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Klinik für Kardiologie, Pneumologie und Angiologie, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: PVI
Record Dates: First submitted 2016-02-18; First posted 2016-04-12 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; pulmonary vein isolation; heart rate turbulence; baroreflex sensitivity
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pulmonary vein isolation (PVI) has become a standard therapy for atrial fibrillation (AF), however, there is still considerable AF recurrence after PVI. Except for PV-left atrium (LA) reconnection, the cause of recurrence has been not yet fully clarified.

The alternation of autonomic tone plays an important role in initiation of paroxysmal AF. It was reported that there are multiple gangliated plexus (GP) around pulmonary veins, therefore the modulation targeting those GPs, resulting in modulations of cardiac autonomic tone, have been conducted. Some study showed the efficacy of GP ablation for AF patients.

According to the previous reports, heart rate (HR) increased, and heart rate variability (HRV) reduced after PVI. These are considered to be due to "autonomic denervation" caused by catheter ablation of GP.

For the best of investigators knowledge, there have been no data on heart rate turbulence (HRT) of baroreflex sensitivity (BRS) concerning PVI.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo PVI for paroxysmal atrial fibrillation
* Patients in sinus rhythm at baseline

Exclusion Criteria:

* prior left atrial Ablation
* left atrial diameter >55mm
* frequent atrial extrasystole, frequent ventricular Extrasystole
* Diabetes Mellitus
* sleep apnea syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo PVI for paroxysmal AF
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
recurrence of AF | 12 months
  Time measured in days to recurrence of AF

SECONDARY OUTCOMES:
effect of PVI on cardiac autonomic system utilizing HRT measurement | 12 months
effect of PVI on cardiac autonomic system utilizing BRS measurement | 12 months
association between measured parameters (HRT, BRS) and the recurrence of AF | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hisaki Makimoto, MD, Principal Investigator — Division of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany